CLINICAL TRIAL: NCT02072720
Title: Pilot Study to Determine the Effect of Fractionated Radiotherapy on Expression of Pro-angiogenic Factors in Oesophagus Carcinoma
Brief Title: Angiogenic Factor Expression During Fractionated Irradiation
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Noordwest Ziekenhuisgroep (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, H.M.W. Verheul, Prof. H.M.W. Verheul, Amsterdam UMC, location VUmc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013/340
Record Dates: First submitted 2014-02-19; First posted 2014-02-26 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Primary Esophageal Carcinoma
Keywords: Radiotherapy; VEGF; esophagus carcinoma; bevacizumab
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- on-treatment tumor biopsie (No Intervention): patients will undergo an pre-treatment and on-treatment tumor biopsy, to measure VEGF expression, and identify the time point of induction of VEGF expression.
- bevacizumab (Experimental): These patients will receive bevacizumab once a week during their chemoradiation, starting at the identified time point of enhanced VEGF expression. These patients will also undergo and pre-treatment tumor biopsy and 1 tumor biopsy 1 week after the start of bevacizumab treatment.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — patients will receive bevacizumab (3mg/kg/wk) starting from the identified induction time point of VEGF expression
  Other Names: Bevacizumab (Avastin).
  Arms: bevacizumab

SUMMARY:
The main question of this study is if and when VEGF (vascular endothelial growth factor) expression in the tumor is upregulated during chemoradiation and if bevacizumab inhibits subsequent vessel growth in the tumor.

* Therefore the first aim of this study is to identify the time point of induction of VEGF in the tumor tissue of esophagus carcinoma during chemoradiation (after 1,2,3 or 4 weeks of chemoradiation).
* If we identify increased expression of VEGF at a certain time point, our second aim is to determine if we can inhibit the subsequent tumor vessel growth by administration of bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* patients that will receive chemoradiation following CROSS-schedule before surgery for esophageal carcinoma
* ability to give informed consent
* age 18 years or older

Exclusion Criteria:

* pregnancy
* evidence of bleeding diathesis, coagulopathy
* inflammation of the GI-tract
* brain metastases
* diastolic/ systolic hypertension, not responding to treatment
* arterial thromboembolism in medical history
* surgery within the month prior to start of bevacizumab treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-02; Primary Completion 2021-03 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Change of VEGF mRNA expression in tumor biopsies | 5 weeks
  To compare the VEGF mRNA expression in the pre-treatment and on-treatment tumor biopsies, to measure the change in VEGF expression from baseline.
Change of VEGFR2 phosphorylation with IHC | 8 weeks
  To determine the level of pVEGFR2 expression in tumor biopsies of patients that received bevacizumab, and to compare that to their pre-treatment expression levels, to identify the changes in expression from baseline.

SECONDARY OUTCOMES:
Changes of mRNA expression of other pro-angiogenic factors | 5 weeks
  To identify the expression of other pro-angiogenic factors in the tumor, and to measure the changes from baseline expression (pre-treatment vs on-treatment biopsies).
Changes in protein expression of pro-angiogenic factors | 5 weeks
  To identify the protein expression of other pro-angiogenic factors in the tumor, and to measure the changes from baseline expression (pre-treatment vs on-treatment biopsies).
Changes in vascular parameters in the tumor tissue to asses ongoing angiogenesis | 5 weeks
  To identify the expression of CD31+ and pericyte markers with IHC staining in the tumor, and to measure the changes from baseline expression (pre-treatment vs on-treatment biopsies).

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - VU university medical center, Amsterdam, North Holland
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Academisch Medisch Centrum, Amsterdam